CLINICAL TRIAL: NCT02998970
Title: Effects of Empagliflozin on Cardiac Structure, Function, and Circulating Biomarkers in Patients With Type 2 Diabetes
Brief Title: Effects of Empagliflozin on Cardiac Structure in Patients With Type 2 Diabetes
Acronym: EMPA-HEART
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: REB# 15-402
Record Dates: First submitted 2016-12-05; First posted 2016-12-21 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Diabetes; Cardiovascular Disease
Keywords: Cardiovascular Disease; Type 2 Diabetes; Cardiac Magnetic Resonance Imaging
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases; Diabetes Mellitus, Type 2 | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): The placebo group acts as a control group. This is in order to objectively isolate empagliflozin's effect on cardiac structure and function as determined by CMR imaging.
  Interventions: Drug: Placebo
- Empagliflozin (Active Comparator): The study medication (Jardiance) is the only diabetes medication to show a significant reduction in both cardiovascular risk and cardiovascular death. The generic name is empagliflozin and will be provided by Boehringer-Ingelheim. If the patient is randomized into the study drug group patients will receive empagliflozin 10 mg tablets once daily for a duration of 6 months.
  Interventions: Drug: Empagliflozin

INTERVENTIONS:
Drug: Empagliflozin — single oral tablet once daily.
  Other Names: Jardiance
  Arms: Empagliflozin
Drug: Placebo — single oral tablet once daily.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effects of Empagliflozin on cardiac structure, function and circulating biomarkers in patients with Type II diabetes. Empagliflozin (anti-hyperglycemic agent), approved by Health Canada and the FDA for the treatment of Type II diabetes, demonstrated a reduction in cardiovascular deaths and heart failure from a previous post-marketing clinical trial. The use of empagliflozin to treat patients with diabetes and heart disease has been approved by Health Canada. However, the process by which it may give this beneficial effect remains unclear and needs further investigation. Therefore, the aim of this study is to provide a fundamental understanding of the mechanistic basis by which Empagliflozin could provide its potential cardio-protective effects by employing the use of Cardiac Magnetic Resonance Imaging (CMRI).

DETAILED DESCRIPTION:
The prevalence of heart failure in Canada is high, affecting 1-3% of total population, representing one of the health care system's most expensive diagnoses. Type 2 diabetes is a significant risk factor for heart disease, and the presence of both type 2 diabetes and heart disease increases the risk of other major health complications including death. A translational study is fundamental in understanding of the potential mechanistic basis of empagliflozin's cardiac benefit.

The study drug, empagliflozin (marketed as Jardiance), belongs to a class of medications that lowers blood glucose (sugar) by preventing glucose from entering back into blood circulation and ensures it is eliminated in urine. It is approved by the FDA and Health Canada for the treatment of type 2 diabetes.

This is a double-blind, randomized, placebo-controlled, parallel-group phase IV study of empagliflozin vs. placebo in patients with type 2 diabetes with inadequate glycemic control and at high cardiovascular risk. The purpose is to better understand how empagliflozin could potentially improve heart function with the use of CMRI. Patients who have given informed consent will undergo a baseline CMRI and will then be randomly assigned in a 1:1 basis to either empagliflozin 10 mg once daily (OD) or matching placebo. The aim of the study is to consent 90 eligible subjects, who will be followed for 26 weeks. An end of study CMRI will be performed at 26 weeks.

The study is comprised of 6 study visits and enrolled subjects will be followed for 6 months. The patients will be assessed using CMRI, which is considered the "gold standard" for measuring left ventricular (LV) volume, mass, and ejection fraction. Patients will undergo two CMRI examinations: at baseline and 6 months after surgery.

In addition, the investigators will be investigating changes from baseline in LV end-diastolic volume, end-systolic volume, LV ejection fraction, regional LV diastolic and systolic function, aortic pulse wave velocity and distensibility (as measures of arterial stiffness) via CMR imaging in patients with type 2 diabetes treated with empagliflozin compared to those who receive placebo. Also, changes from baseline on a panel of biomarkers involved in the pathophysiology of heart will be evaluated at baseline, 1 months and 6 months, in patients with type 2 diabetes treated with empagliflozin.

Study assessments and potential adverse events reporting will be undertaken at each study visit.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ≥40 and ≤ 80 years of age
* History of type 2 diabetes
* Haemoglobin A1C ≥6.5 and ≤10 % within 3 months of the Screening Visit
* Established cardiovascular disease, defined as previous myocardial infarction ≥ 6 months ago, or previous coronary revascularization ≥ 2 months ago
* Any background antihyperglycemic therapy (which has been stable for at least 2 months)
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the trial
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests and other trial procedures

Exclusion Criteria:

* Female subjects who are pregnant, lactating or of child bearing potential, or pre-menopausal women. (Menopause will be determined by patient and physician history)
* Type 1 diabetes
* Subjects currently treated with SGLT2 inhibitors, Glucagon-like peptide-1 (GLP1) receptor agonist, or saxagliptin
* Frequent episodes (>4/month) of moderate hypoglycaemia, as defined by the Canadian Diabetes Association 2013 Clinical Practice Guidelines for the Prevention and Management of Diabetes
* Any episode of severe hypoglycaemia within the past 12 months, as also defined by the Canadian Diabetes Association 2013 Clinical Practice Guidelines for the Prevention and Management of Diabetes
* Subjects in whom coronary revascularisation by either Percutaneous coronary intervention (PCI) or bypass surgery is being contemplated within 6 months, or who have undergone revascularisation in the prior 2 months
* Modification of Diet in Renal Disease (MDRD) Estimated Glomerular Filtration Rate (eGFR)< 60 ml/min/1.73 m2 at screening
* Significant allergy or known intolerance to SGLT2 inhibitors or any ingredient in the formulations
* Subjects currently experiencing any clinically significant or unstable medical condition that might limit their ability to complete the study, or to comply with the requirements of the protocol, including: dermatologic disease, haematological disease, pulmonary disease, hepatic disease, gastrointestinal disease, genitourinary disease, endocrine disease, neurological disease and psychiatric disease
* Any malignancy not considered cured (except basal cell carcinoma of the skin). A subject is considered cured if there has been no evidence of cancer recurrence for the 5 years prior to screening
* Blood donation within 4 weeks prior to screening, or stated intention to donate blood or blood products during the period of the study or within one month following completion of the study
* Subjects who have participated in studies of an investigational drug or device within 30 days prior to the screening visit
* Conditions preventing safe MRI imaging such as the subject's weight exceeding 500 lbs; maximum body dimension from side-to-side exceeding 70 cm and from back to front of torso exceeding 50 cm or the presence of metallic fragments, clips or devices
* LVEF <30% on the most recent assessment within 6 months
* New York Heart Association (NYHA) Class IV or recent hospitalization for decompensated Heart Failure (HF) (<3 months)
* Unstable coronary syndromes
* Moderate or severe aortic stenosis
* Moderate or severe aortic regurgitation
* Moderate or severe mitral stenosis
* Moderate or severe mitral regurgitation

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Left Ventricular (LV) mass Changes | 6 months
  Changes in Left Ventricular (LV) mass (indexed to BSA) at 6 months in patients with Type 2 diabetes who receive empagliflozin vs. placebo.
  This will be measured using CMRI.

SECONDARY OUTCOMES:
LV end-diastolic volume | 6 months
  Changes in LV end-diastolic volume (indexed to BSA) at baseline and at 6 months in patients with type 2 diabetes treated with empagliflozin.
  This will be measured using CMRI.
End-systolic volume (indexed to BSA) | 6 months
  Changes in end-systolic volume (indexed to BSA) at baseline and at 6 months in patients with type 2 diabetes treated with empagliflozin.
  This will be measured using CMRI.
Left Ventricular Ejection Fraction (LVEF) | 6 months
  Changes LVEF at baseline and at 6 months in patients with type 2 diabetes treated with empagliflozin.
  This will be measured using CMRI.
Regional LV diastolic function | 6 months
  Changes in Regional LV diastolic function at baseline and at 6 months in patients with type 2 diabetes treated with empagliflozin.
  This will be measured using CMRI.
Regional LV systolic function | 6 months
  Changes in Regional LV systolic function at baseline and at 6 months in patients with type 2 diabetes treated with empagliflozin.
  This will be measured using CMRI.
Aortic pulse wave velocity and distensibility | 6 months
  Changes in aortic pulse wave velocity and distensibility (as arterial stiffness) at baseline and at 6 months in patients with type 2 diabetes treated with empagliflozin.
Biomarkers | 6 months
  Changes on a panel of biomarkers involved in the pathophysiology of heart failure at baseline, 1 months and 6 months, in patients with type 2 diabetes treated with empagliflozin.
Plasma catecholamine levels | 6 months
  Changes in plasma catecholamine levels at baseline, 1 months and 6 months, in patients with type 2 diabetes treated with empagliflozin.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pourafkari M, Connelly KA, Verma S, Mazer CD, Teoh H, Quan A, Goodman SG, Rai A, Ng MY, Deva DP, Triverio P, Jiminez-Juan L, Yan AT, Ge Y. Empagliflozin and left atrial function in patients with type 2 diabetes mellitus and coronary artery disease: insight from the EMPA-HEART CardioLink-6 randomized clinical trial. Cardiovasc Diabetol. 2024 Aug 28;23(1):319. doi: 10.1186/s12933-024-02344-6. PMID 39198860
- [Derived] Barbour W, Wolff E, Puar P, Hibino M, Bakbak E, Krishnaraj A, Verma R, Verma M, Quan A, Yan AT, Connelly KA, Teoh H, Mazer CD, Verma S. Effect of empagliflozin on cardiac remodelling in South Asian and non-South Asian individuals: insights from the EMPA-HEART CardioLink-6 randomised clinical trial. BMC Cardiovasc Disord. 2023 Nov 15;23(1):557. doi: 10.1186/s12872-023-03549-5. PMID 37964221
- [Derived] Puar P, Ahmed S, Hibino M, Pasricha A, Pandey A, Bari A, Verma R, Quan A, Yan AT, Connelly KA, Teoh H, Mazer CD, Verma S. The association between anthropometric indicators of obesity and cardiac reverse remodelling with empagliflozin in patients with type 2 diabetes and coronary artery disease. Diabetes Obes Metab. 2023 Sep;25(9):2765-2769. doi: 10.1111/dom.15119. Epub 2023 May 29. No abstract available. PMID 37246798
- [Derived] Sarak B, Verma S, David Mazer C, Teoh H, Quan A, Gilbert RE, Goodman SG, Bami K, Coelho-Filho OR, Ahooja V, Deva DP, Garg V, Gandhi S, Connelly KA, Yan AT. Impact of empagliflozin on right ventricular parameters and function among patients with type 2 diabetes. Cardiovasc Diabetol. 2021 Oct 4;20(1):200. doi: 10.1186/s12933-021-01390-8. PMID 34607574
- [Derived] Mason T, Coelho-Filho OR, Verma S, Chowdhury B, Zuo F, Quan A, Thorpe KE, Bonneau C, Teoh H, Gilbert RE, Leiter LA, Juni P, Zinman B, Jerosch-Herold M, Mazer CD, Yan AT, Connelly KA. Empagliflozin Reduces Myocardial Extracellular Volume in Patients With Type 2 Diabetes and Coronary Artery Disease. JACC Cardiovasc Imaging. 2021 Jun;14(6):1164-1173. doi: 10.1016/j.jcmg.2020.10.017. Epub 2021 Jan 13. PMID 33454272
- [Derived] Verma S, Mazer CD, Yan AT, Mason T, Garg V, Teoh H, Zuo F, Quan A, Farkouh ME, Fitchett DH, Goodman SG, Goldenberg RM, Al-Omran M, Gilbert RE, Bhatt DL, Leiter LA, Juni P, Zinman B, Connelly KA. Effect of Empagliflozin on Left Ventricular Mass in Patients With Type 2 Diabetes Mellitus and Coronary Artery Disease: The EMPA-HEART CardioLink-6 Randomized Clinical Trial. Circulation. 2019 Nov 19;140(21):1693-1702. doi: 10.1161/CIRCULATIONAHA.119.042375. Epub 2019 Aug 22. PMID 31434508